CLINICAL TRIAL: NCT06868862
Title: Acute Physiological Responses to Isoenergetic High-Intensity Interval Vs. Moderate-Intensity Continuous Exercise in Overweight or Obese Young Females: Focus on Catecholamines, Oxygen Consumption, Lipid Utilization, and Appetite Regulation
Brief Title: Acute Effects of Isoenergetic HIIE Vs. MICE on Key Parameters of Fat Mass Loss in Young Females with Overweight or Obesity
Acronym: COMEFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Collaborators: LAPEF laboratory, Sao paulo (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE: 79561024.4.0000.9487
Record Dates: First submitted 2025-02-21; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obese Adults; High Intensity Interval Exercise (HIIE)
Keywords: oxygen consumption; high intensity interval training; substrate oxydation; catecholamines; obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data collected on the volunteers will be made anonymous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Interval Exercise (Experimental): High Intensity Interval Exercise: 5 minutes of WarmUp + 10 x (1 minute at 85% HRmax followed by 1 minute of recovery at a power equivalent to 40% of HRmax)
  Interventions: Other: Exercise
- Moderate Intensity Continuous Exercise (Experimental): Moderate Intensity Continuous Exercise: 5 minutes of WarmUp + 35 minutes at 55% HRmax
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Two Exercise Modalities: HIIE and MICE

SUMMARY:
Overweight and obesity, particularly increased total and/or abdominal fat mass (FM), are strongly linked to the development of cardiovascular diseases. Managing obesity effectively requires lifestyle and dietary modifications, including increased physical activity. Among the various exercise strategies, Moderate-Intensity Continuous Training (MICT) and High-Intensity Interval Training (HIIT) are widely recommended for reducing FM. Compared to MICT, HIIT is a time-efficient approach, often perceived as more enjoyable, and has been shown to promote greater total and abdominal fat loss in a shorter period. However, the precise mechanisms underlying this enhanced fat loss remain unclear.

This study aims to compare the acute effects of two isoenergetic exercise sessions - MICE (Moderate-Intensity Continuous Exercise) and HIIE (High-Intensity Interval Exercise) - on key physiological responses involved in fat mass loss. Specifically, we will assess plasma catecholamine levels during exercise and recovery, as well as oxygen consumption, substrate oxidation, and appetite over the 2-hour post-exercise period in young females with overweight or obesity. By elucidating the role of catecholaminergic stimulation as a potential regulator of fat mass loss, this research could provide valuable insights for optimizing exercise strategies in weight management and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* women with overwieght or obesity (BMI: 25-35 kg/m²)

Exclusion Criteria:

* contraceptive use
* menopause
* irregular menstrual cycle
* medical contraindications to intense physical activity,
* painful joints,
* taking ß-blocker

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption during exercise and the recovery period | Measurement at rest for 20 minutes, then during warm-up for 10 minutes, then during exercise for 20 minutes and finally during 2 hours after the end of the exercise.
  Determination of oxygen consumption during exercise and 2 hours after the exercise session (HIIE and MICE). Determination from Metamax (3D Cortex).

SECONDARY OUTCOMES:
Lipid before and after the exercise. | Measurement at rest for 20 minutes and then during 2 hours after the end of the exercise.
  Determination of lipid oxidation before and after the exercise. Lipid oxidation is measured from oxygen and carbon dioxide consumption (Metamax 3D Cortex).
Carbohydrate before and after the exercise. | Measurement at rest for 20 minutes and then during 2 hours after the end of the exercise.
  Determination of carbohydrate oxidation before and after the exercise. Carbohydrate oxidation is measured from oxygen and carbon dioxide consumption (Metamax 3D Cortex).
Catecholamines | 5 collections: before exercise started, at the end of exercise (exercise duration is 20-35 minutes), at 30 minutes, 60 minutes and 120 minutes after the end of exercise
  Determination of cathecolamines concentration in blood during exercise and 2 hours after the end of the exercise.
Energy intakes 24 hours after the exercise | 24 hours post exercise
  Evaluation of energy intakes after the exercise session (HIIE vs MICE). Exercise session finish at 11:30 a.m. After that, at home, participants have to complete by themselves a food-record on which they will describe all their meal during 24 hours after the end of the exercise session. It includes their lunch, dinner and their breakfast the next morning.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Fisiologia e Metabolismo Aplicados à Educação Física, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dupuit M, Rance M, Morel C, Bouillon P, Pereira B, Bonnet A, Maillard F, Duclos M, Boisseau N. Moderate-Intensity Continuous Training or High-Intensity Interval Training with or without Resistance Training for Altering Body Composition in Postmenopausal Women. Med Sci Sports Exerc. 2020 Mar;52(3):736-745. doi: 10.1249/MSS.0000000000002162. PMID 31524825
- [Background] Dupuit M, Boscaro A, Bonnet A, Bouillon P, Bruno P, Morel C, Rance M, Boisseau N. Acute metabolic responses after continuous or interval exercise in post-menopausal women with overweight or obesity. Scand J Med Sci Sports. 2020 Dec;30(12):2352-2363. doi: 10.1111/sms.13814. Epub 2020 Sep 18. PMID 32881054
- [Background] Cunha FA, Midgley AW, McNaughton LR, Farinatti PT. Effect of continuous and intermittent bouts of isocaloric cycling and running exercise on excess postexercise oxygen consumption. J Sci Med Sport. 2016 Feb;19(2):187-92. doi: 10.1016/j.jsams.2015.02.004. Epub 2015 Feb 23. PMID 25747467